CLINICAL TRIAL: NCT05116839
Title: Pressure Support Ventilation Versus Continuous Positive Air Way Pressure (CPAP) Using I Gel Laryngeal Mask for Minor Surgery in Adult Patients, a Prospective cross_over Study
Brief Title: Pressure Support Ventilation Versus Continuous Positive Air Way Pressure (CPAP) Using I Gelin Adult Patients,
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Marwa Ibrahim Mohamed Abdo,MD, Lecturer of Anesthesia and Surgical Intensive Care-Faculty of Medicine - Mansoura University, Mansoura University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: MS/19.03.556
Record Dates: First submitted 2021-08-20; First posted 2021-11-11 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Ventilator Lung
Keywords: Pressure support ventilation (CPAP) I gel
MeSH Terms: conditions — Microcephaly, Primary Autosomal Recessive, 6

STUDY DESIGN:
Intervention Model Description: a prospective cross_over study
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the first 15 minutes with PSV (Placebo Comparator): All patients will breath at the first 15 minutes with PSV:triggered by minute volume <3 Liter,with with no frequency .
  Monitoring: (basal&every 3minutes)
  1. Tidal volume (inspiratory & expiratory).
  2. End tidal co2.
  3. Mean air way pressure.
  4. Leakage %.
  5. Respiratory rate .
  6. Spo2.
  7. Heart rate.
  8. Blood pressure (mean arterial pressure
  Interventions: Device: the first 15 minutes with pressure support ventilation; Device: i gel air way
- the following 15 minutes ventilation will be changed to CPAP mode (Active Comparator): then the following 15 minutes ventilation will be changed to CPAP mode at 10 cm H2o .
  Monitoring: (basal&every 3minutes)
  1. Tidal volume (inspiratory & expiratory).
  2. End tidal co2.
  3. Mean air way pressure.
  4. Leakage %.
  5. Respiratory rate .
  6. Spo2.
  7. Heart rate.
  8. Blood pressure (mean arterial pressure).
  Interventions: Device: the following 15 minutes ventilation will be changed to continous positive air way pressureCPAP mode; Device: i gel air way

INTERVENTIONS:
Device: the first 15 minutes with pressure support ventilation — PSV pressure support ventilation:triggered by minute volume < 3 Liter ,with no frequency
  Other Names: lung mechanical ventilatory mode on mechanical ventilator
  Arms: the first 15 minutes with PSV
Device: the following 15 minutes ventilation will be changed to continous positive air way pressureCPAP mode — continous positive air way pressure CPAP mode at 10 cm H2o .
  Other Names: lung mechanical ventilatory mode on mechanical ventilator
  Arms: the following 15 minutes ventilation will be changed to CPAP mode
Device: i gel air way — supraglottic air way device

SUMMARY:
Introduction of Supra glottic airway devices (SAD) has revolutionized the airway management. The first successful supraglottic airway device, the Laryngeal Mask Airway(LMA).The various other SADs include ProSeal LMA, Intubating LMA and i-gel to overcome the limitations of classic Laryngeal Mask Airway( c-LMA) The risk of aspiration with c-LMA is reported tobe around 9% , pleaseboth the c-LMA and PLMA have cuff related complications. High cuff pressure in laryngeal mask airways can cause damage to the mucosae on periglottic and supraglottic structures .

Therefore, to overcome the limitations of Pro Seal Laryngeal Mask Airway (PLMA )a new and cheaper SAD called i-gel was developed. i-gel is a novel and innovative, latex free supraglottic device, made up of medical grade thermoplastic elastomer, which is soft, gel like, transparent The number of manipulations required are more in PLMA than i gel resulting in hemodynamic changes .The i-gel is comparable to PLMA insuring the airway during controlled ventilation. It is better than PLMA in terms of ease of insertion.

Spontaneous breathing is the most popular mode of ventilation with the laryngeal mask airway (LMA), but it provides less effective gas exchange than does positive pressure ventilation (PPV) . The patients receiving sevoflurane anesthesia with unassisted ventilation have a reduced rib cage contribution to ventilation, decreased tidal volume, and respiratory rate .

Pressure support ventilation (PSV) is a ventilator mode that is initiated by the patient and synchronized with the patient's respiratory effort. And may improve gaseous exchange in patients. In the intensive care unit, it is often considered the preferred mode for weaning mechanical ventilation .PSV provides more effective gas exchange than does unassisted ventilation with CPAP during anesthesia with the LMA while preserving hemodynamic homeostasis.

The use of PSV versus CPAP with the Pro Seal laryngeal mask airway in anesthetized pediatric patients revealed that PSV improved gaseous exchange and reduced work of breathing during general anesthesia PSV via Pro- Seal laryngeal mask airway improves gaseous exchange and ventilation in pediatric patients under general anesthesia more than spontaneous ventilation .

DETAILED DESCRIPTION:
Patients and Methods This prospective,cross over study will be conducted after obtaining approval from the Institutional Review Board (IRB) of faculty of medicine Mansoura University. A written informed consent will be obtained from all participants and the duration of the study will be 2 - 6 months.

Participants:

38 Adult patients with American Society of Anesthesiologists (ASA) physical status (I - II )of both sexes aged (18-65) years scheduled for minor surgery at Urology and Nephrology centre (UNC) will be included in this study.

The Patients with a body mass index (BMI) >40 or having obstructive air way disease will be excluded.

All patients will be assessed on the day before surgery by detailed history thorough clinical examination, and basal laboratory investigations [Complete blood count (CBC), Coagulation profile (prothrombin time and INR), liver and renal function tests (liver enzymes, bilirubin, albumin and s. creatinine], electrocardiograph (ECG) and echo cardiography when needed.

Anaesthesia Induction of anaesthesia with fentanyl 0.5µg/kg - propofol 1mg/kg prior for insertion of device,primary success rate will be recorded.

Maintenance of anaesthesia by sevoflurane inhalation with minimal alveolar concentration (MAC) 2%.

All patients will breath spontaneously from ventilators (Dragers - Primal - germany).

All patients will breath at the first 15 minutes with PSV:triggered by minute volume <3 liter,with no frequency then the following 15 minutes ventilation will be changed to CPAP mode at 10 cm H2o .

Monitoring: (basal& every 3minutes)

1. Tidal volume (inspiratory & expiratory).
2. End tidal co2.
3. Mean air way pressure.
4. Leakage %.
5. Respiratory rate .
6. Spo2.
7. Heart rate.
8. Blood pressure (mean arterial pressure). Adverse effects;Laryngeal spasm.Blood stained device. .

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with (ASA) physical status I - II years scheduled for minor surgery at Urology and Nephrology centre (UNC) will be included in this study.

Exclusion Criteria:

* The Patients with a body mass index (BMI) >40 or having obstructive air way disease will be excluded.•

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2019-03-31 (Actual); Primary Completion 2021-12-28 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
Effective ventilation with PSV than does (CPAP) as regard Tidal volume | 30 minutes
  Breathing of all patients at the first 15 minutes with PSV pressure support ventilation:triggered by minute volume <3 liter,with no frequency then the following 15 minutes ventilation with CPAP .ventilation will be measured by Monitoring: (basal& every 3minutes)Tidal volume (inspiratory & expiratory).on ventilator monitor in mil/ kilogram
Effective ventilation with PSV than does (CPAP) as regard End tidal co2. on ventilator | 30 minutes
  Breathing of all patients at the first 15 minutes with PSV pressure support ventilation:triggered by minute volume <3 liter,with no frequency then the following 15 minutes ventilation with CPAP.ventilation will be measured by Monitoring: (basal& every 3minutes) End tidal co2. on ventilator ml/eq
Effective ventilation with PSV than does CPAP as regard Mean air way pressure | 30 minutes
  Breathing of all patients at the first 15 minutes with PSV pressure support ventilation:triggered by minute volume <3 liter,with no frequency then the following 15 minutes ventilation with CPAP.ventilation will be measured by Monitoring: (basal& every 3minutes) Mean air way pressure.on ventilator mmhg
Effective ventilation with PSV than does (CPAP) as regard Leakage % | 30 minutes
  Breathing of all patients at the first 15 minutes with PSVpressure support ventilation:triggered by minute volume <3 liter,with no frequency then the following 15 minutes ventilation with CPAP.ventilation will be measured by Monitoring: (basal& every 3minutes) Leakage % on ventilator monitor
Effective ventilation with PSV than does CPAP as regard oxygen saturation. | 30 minutes
  Breathing of all patients at the first 15 minutes with PSV pressure support ventilation:triggered by minute volume <3 liter,with no frequency then the following 15 minutes ventilation with CPAP.ventilation will be measured by Monitoring: (basal& every 3minutes) oxygen saturation.on monitoring in %
Effective ventilation with PSV than does (CPAP) as regard respiratory rate | 30 minutes
  Breathing of all patients at the first 15 minutes with PSV pressure support ventilation:triggered by minute volume <3 liter,with no frequency then the following 15 minutes ventilation with CPAP .ventilation will be measured by Monitoring: (basal& every 3minute)respiratory rate on monitor breath/ minute

CONTACTS AND LOCATIONS:
Overall Officials: Golnar Se Hammouda, M.D, Study Chair — Professor of Anesthesia Intensive Care Faculty of Medicine - Mansoura University; Hanaa Ma El-Bendary, M.D, Study Director — Assistant Professor of Anesthesia Intensive Care Faculty of Medicine - Mansoura University; Marwa Ib Abdo, M.D, Principal Investigator — Lecturer of Anesthesia Intensive Care Faculty of Medicine - Mansoura University; Bahaa Mo Ezz, MBBCh, Principal Investigator — Resident of Anesthesia Intensive Care Mansoura University Hospitals
Locations (1):
- Marwa Ibrahim Mohamed abdo, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barker P, Langton JA, Murphy PJ, Rowbotham DJ. Regurgitation of gastric contents during general anaesthesia using the laryngeal mask airway. Br J Anaesth. 1992 Sep;69(3):314-5. doi: 10.1093/bja/69.3.314. PMID 1389850
- [Background] Wong JG, Heaney M, Chambers NA, Erb TO, von Ungern-Sternberg BS. Impact of laryngeal mask airway cuff pressures on the incidence of sore throat in children. Paediatr Anaesth. 2009 May;19(5):464-9. doi: 10.1111/j.1460-9592.2009.02968.x. Epub 2009 Mar 5. PMID 19281479
- [Background] Levitan RM, Kinkle WC. Initial anatomic investigations of the I-gel airway: a novel supraglottic airway without inflatable cuff. Anaesthesia. 2005 Oct;60(10):1022-6. doi: 10.1111/j.1365-2044.2005.04258.x. PMID 16179048
- [Background] Chauhan G, Nayar P, Seth A, Gupta K, Panwar M, Agrawal N. Comparison of clinical performance of the I-gel with LMA proseal. J Anaesthesiol Clin Pharmacol. 2013 Jan;29(1):56-60. doi: 10.4103/0970-9185.105798. PMID 23493414
- [Background] Verghese C, Brimacombe JR. Survey of laryngeal mask airway usage in 11,910 patients: safety and efficacy for conventional and nonconventional usage. Anesth Analg. 1996 Jan;82(1):129-33. doi: 10.1097/00000539-199601000-00023. PMID 8712387
- [Background] Keller C, Sparr HJ, Luger TJ, Brimacombe J. Patient outcomes with positive pressure versus spontaneous ventilation in non-paralysed adults with the laryngeal mask. Can J Anaesth. 1998 Jun;45(6):564-7. doi: 10.1007/BF03012709. PMID 9669012
- [Background] Tokioka H, Nagano O, Ohta Y, Hirakawa M. Pressure support ventilation augments spontaneous breathing with improved thoracoabdominal synchrony in neonates with congenital heart disease. Anesth Analg. 1997 Oct;85(4):789-93. doi: 10.1097/00000539-199710000-00013. PMID 9322456
- [Background] Farias JA, Frutos F, Esteban A, Flores JC, Retta A, Baltodano A, Alia I, Hatzis T, Olazarri F, Petros A, Johnson M. What is the daily practice of mechanical ventilation in pediatric intensive care units? A multicenter study. Intensive Care Med. 2004 May;30(5):918-25. doi: 10.1007/s00134-004-2225-5. Epub 2004 Mar 17. PMID 15029473
- [Background] Brimacombe J, Keller C, Hormann C. Pressure support ventilation versus continuous positive airway pressure with the laryngeal mask airway: a randomized crossover study of anesthetized adult patients. Anesthesiology. 2000 Jun;92(6):1621-3. doi: 10.1097/00000542-200006000-00019. PMID 10839911
- [Background] von Goedecke A, Brimacombe J, Hormann C, Jeske H-, Kleinsasser A, Keller C. Pressure support ventilation versus continuous positive airway pressure ventilation with the ProSeal laryngeal mask airway: a randomized crossover study of anesthetized pediatric patients. Anesth Analg. 2005 Feb;100(2):357-360. doi: 10.1213/01.ANE.0000143563.39519.FD. PMID 15673856
- [Background] Lim B, Pawar D, Ng O. Pressure support ventilation vs spontaneous ventilation via ProSeal laryngeal mask airway in pediatric patients undergoing ambulatory surgery: a randomized controlled trial. Paediatr Anaesth. 2012 Apr;22(4):360-4. doi: 10.1111/j.1460-9592.2012.03819.x. PMID 22380745